CLINICAL TRIAL: NCT06779760
Title: Assessing the Feasibility of Near Infrared Autofluorescence Imaging in Minimally-Invasive Video-Assisted Parathyroidectomy and the Autofluorescence Signature of Parathyroid Adenomas
Brief Title: Near Infrared Autofluorescence Imaging in Minimally-Invasive Video-Assisted Parathyroidectomy (NIRAF MIVAP Study)
Acronym: NIRAF MIVAP
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: The Hashemite University (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Professor of Surgery, Aristotle University Of Thessaloniki
Other Study IDs: NIRAF MIVAP study
Record Dates: First submitted 2024-11-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: Primary Hyperparathyroidism Due to Adenoma
Keywords: primary hyperparathyroidism; parathyroid adenoma; near-infrared autofluorescence; minimally invasive parathyroidectomy
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism, Primary | interventions — Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: parathyroidectomy — The FLUOBEAM® LX apparatus consists of a camera with a built-in light emitter (750-800 nm) and detector (800-830 nm) connected to a processor with an indication-oriented software (Fluosoft®). The processor captures the emitted light, allowing display of PTG images in real time. The camera is placed in a sterile sheath and is held perpendicularly at 8 cm from the target tissue with operating lights, all background lights, and any ambient light being extinguished. The reported depth of tissue penetration of near-infrared light is limited to a maximum of 3 mm only with no observed differences between superior and inferior PTGs [10]. This highlights the importance of a major surgical technical point "reaching the correct plane of dissection" namely, the pre-vertebral fascia to maximize the chances of eliciting an adequate signal from parathyroid tissue. The correct application of the technology has demonstrated a success rate of signal elicitation of 90%-100% [11]. The ability of near-infr

SUMMARY:
The role of near-infrared autofluorescence (NIRAF)-imaging as an adjunct in thyroid surgery is well established. However, its diagnostic role in hyperparathyroidism surgery is yet to be defined due to the lack of consensus regarding the autofluorescence (AF) pattern of pathological parathyroid glands. Furthermore, its utility via a direct minimal access has not been assessed.

To assess the AF pattern of parathyroid adenomas (PAs) utilizing NIRAF-imaging in minimally invasive video-assisted parathyroidectomy (MIVAP).

The clinical records of patients who underwent MIVAP for hyperparathyroidism between February and October 2024 were retrospectively reviewed. The primary endpoint was to assess the AF pattern of PAs. Secondary endpoints included the feasibility of applying NIRAF imaging in MIVAP and whether certain AF patterns of PAs correlated with cell type, size, and/or location. Furthermore, operative-time and cost implications were assessed.

DETAILED DESCRIPTION:
Native fluorescence or autofluorescence (AF) is defined as the emission of light by a naturally occurring fluorophore, on excitation by incident light of a specific wavelength. Accordingly, fluorescence produced by an endogenous fluorophore differs from that resulting from the application of a synthetic fluorescent marker and is, therefore, considered "contrast-free fluorescence." Maximal AF from both thyroid and parathyroid tissue occurs at the near-infrared spectrum (820-830 nm wavelength) with parathyroid tissue maximal emission intensity being 2-20 times greater than that of thyroid tissue and lasts at least for one hour in vivo. This is probably attributed to that the fluorophore assumed to be responsible for thyroid and parathyroid tissue AF is the calcium-sensing receptor that is present in parafollicular cells (C-cells), but to a much higher extent in parathyroid tissue. This allows for PTGs to be visualized as bright spots on a background of low fluorescence (thyroid gland). The fact that AF persists for at least an hour even after gland devascularization or unintentional resection, implies that NIRAF cannot confirm PTG viability. Viability depends on adequate tissue perfusion. This in turn requires assessing tissue vascularity using AF from a synthetic fluorescent marker such as indocyanine green (ICG); the concept of contrast-enhanced AF rather than contrast-free AF.

The property of AF in a tissue depends on the concentration of the endogenous fluorophore and whether it is affected by a pathological process. Hence, its application in clinical practice allowing it to serve as an optical biopsy (a point detection tool that provides real-time, non-invasive diagnostic information without physically exciting tissue). This might explain why unlike normal parathyroid tissue, parathyroid adenomas (PAs) demonstrate a heterogenous pattern of AF. Demarchi et al. reported that most PAs in their study appeared significantly less autofluorescent than the rim of compressed normal parathyroid tissue (at the periphery of a PA) that appeared as bright cap. This was referred to as cap AF. Nevertheless, no noticeable differences in the pattern of AF between adenomatous, hyperplastic, and normal PTGs were observed by others.

Minimally invasive video-assisted parathyroidectomy (MIVAP) is one of the most popular targeted parathyroid procedures performed for primary hyperparathyroidism. It has been demonstrated that the advantages offered by MIVAP enables it to overcome the limitations of other targeted parathyroid procedures. Allowing for full neck exploration and/or performing a concomitant thyroid procedure without the need to convert to a standard cervicotomy.

The objective of this study was to assess the feasibility of applying NIRAF-imaging via a limited direct access and the potential patterns of AF (AF signature) of PAs on contrast-free NIRAF-based imaging, and whether specific patterns of AF correlated with factors intrinsic to PAs such as the dominant cell type of a PA, its size and/or location. The additional operative time, and cost conferred using this technology were also evaluated

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with parathyroid adenoma undergoing surgery

Exclusion Criteria:

* patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with parathyroid adenoma undergoing surgery and age >18 years old
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
patterns of autofluorescence in parathyroid adenomas | during surgery

SECONDARY OUTCOMES:
specific autofluorescence patterns correlated with the dominant cell type of a parathyroid adenoma | during surgery
specific autofluorescence patterns correlated with adenoma size | during surgery
specific autofluorescence patterns correlated with adenoma location | during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the Hashemite Univesity, Zarqa, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bakkar S, Chorti A, Papavramidis T, Donatini G, Miccoli P. Assessing the feasibility of near infrared autofluorescence imaging in minimally-invasive video assisted parathyroidectomy and the autofluorescence signature of parathyroid adenomas. A single center surgical case series. Surg Endosc. 2025 May;39(5):2964-2972. doi: 10.1007/s00464-025-11675-8. Epub 2025 Mar 21. PMID 40119064